CLINICAL TRIAL: NCT00200850
Title: Sublingual Immunotherapy in Dust Mite Allergy
Brief Title: Immunotherapy Administered Under the Tongue to Treat Dust Mite Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2005-0193; R21AT002326-01A1 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: Breathing; Allergy; Mites, House Dust
MeSH Terms: conditions — Asthma; Respiratory Aspiration; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose SLIT (Active Comparator): Low dose SLIT
  Interventions: Biological: House Dust Mite SLIT
- High dose SLIT (Active Comparator): High dose SLIT
  Interventions: Biological: High dose SLIT
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo SLIT

INTERVENTIONS:
Biological: House Dust Mite SLIT — low dose SLIT 143 Allergen Units(AU)/ml daily
  Arms: Low dose SLIT
Biological: High dose SLIT — House Dust Mite SLIT- 10,000 Allergen units(AU)/ml daily
  Arms: High dose SLIT
Biological: Placebo SLIT — Placebo SLIT daily
  Arms: Placebo

SUMMARY:
This study will investigate sublingual immunotherapy (SLIT), a treatment involving antigens placement under the tongue to help asthma sufferers build a tolerance to the allergy-causing substances. Specifically, this study will determine the effectiveness of SLIT at two different dosing regimens for patients with intermittent mild asthma caused by dust mites.

DETAILED DESCRIPTION:
Asthma is a serious lung condition that is the leading cause of long-term illness in children. Many common household substances can trigger or worsen an asthma attack. It is important for people to reduce household allergens and learn effective treatments for specific types of asthma. Inhaled short-acting beta agonist such as albuterol is the standard treatment for mild, intermittent asthma. However, recent studies have shown that adding allergen-specific immunotherapy to your current asthma therapy can help to control asthma symptoms. This study will determine the safety and effectiveness of SLIT in two different dosing regimens in treating patients with house dust mite-induced allergic rhinitis/mild intermittent asthma.

Participants will be randomly assigned to receive low dose SLIT, high dose SLIT, or placebo for at least 12 months. House dsut mite-induced allergy skin tests will be performed at study entry, at selected timepoints throughout the study, and at the end of the study. The tests will determine whether SLIT creates an immune tolerance state as well as whether SLIT acts via local or systemic immunological systems.

ELIGIBILITY:
Inclusion Criteria:

* House dust mite-induced allergic rhinitis/mild intermittent asthma

Exclusion Criteria:

* Use of previous allergy immunotherapy for house dust mite asthma
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert K. Bush, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin Medical School, Madison, Wisconsin, United States

REFERENCES:
- [Result] Bush RK, Swenson C, Fahlberg B, Evans MD, Esch R, Morris M, Busse WW. House dust mite sublingual immunotherapy: results of a US trial. J Allergy Clin Immunol. 2011 Apr;127(4):974-81.e1-7. doi: 10.1016/j.jaci.2010.11.045. Epub 2011 Feb 18. PMID 21333346

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 31 participants enrolled, 6 participants withdrew due to non-treatment-ascribed-event, 4 participants withdrew due to treatment-ascribed-events.
  Only 21 participants completed the study.
Groups:
- Low Dose: Low dose SLIT
  Hose Dust Mite SLIT: low dose SLIT 143 AU/ml daily
- High Dose: High dose SLIT
  High dose SLIT: House Dust Mite SLIT- 10,000 AU/ml daily
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 10 | 10 | 11
Completed | 7 | 9 | 5
Not Completed | 3 | 1 | 6
Not completed — relocation | 1 | 0 | 1
Not completed — too busy | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Poor adherence | 0 | 0 | 1
Not completed — optic neuritis | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.088) | 33.8 (7.359) | 29.3 (8.634) | 30.6 (7.559)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 8 | 22
  Male | 5 | 1 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 8 | 10 | 11 | 29
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bronchial Threshold to Allergen Challenge From Baseline to 12-18 Months of Treatment
Description: Antigen challenge was performed using the antigen house dust mite. Increasing doses of antigen were inhaled and then lung function (using the procedure Spirometry, measuring Forced Expiatory Volume in the 1st second FEV1) was measured after each dose. The challenge was stopped once the lung function (FEV1) was dropped by 20% of percent predicted. The dose of antigen that caused a 20% drop in lung function is considered the bronchial threshold. The higher the dose of antigen that causes the drop in lung function, the higher tolerance a participant has of inhaling house dust mite. This dose was measure at baseline and then again after 12-18 months of treatment with sublingual house dust mite antigen.Cumulative breath units is the unit of measure to indicate how much antigen is tolerated before the FEV1 is dropped by 20%. Cumulative breath units is also known as breath units.
Time Frame: baseline and after 12-18 months treatment
Measure: Mean (Standard Deviation); unit: cumulative breath units
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 7 | 9 | 5
cumulative breath units
  Baseline dose of antigen | 75.0 (56.7) | 69.5 (46.8) | 141.4 (147)
  Post treatment dose of antigen | 74.8 (57.3) | 100.9 (35.2) | 83.3 (59.3)

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Low Dose | High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=10) | High Dose (N=10) | Placebo (N=11)
oral lesion (General disorders) | 2 (2) | 1 (3) | 4 (5) — Oral lesion or canker sore
throat irritation (General disorders) | 1 (1) | 2 (3) | 1 (1) — Sore throat or strep throat
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 7 (17) | 6 (9) — URI and/or asthma symptoms, pueumonia
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal issues (Gastrointestinal disorders) | 3 (3) | 3 (5) | 1 (1) — Constipation, black stool, nausea
Flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (3)
Head cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (2) | 1 (1) | 1 (1)
Sprain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (6) | 4 (4) — hand wrist, ankle or back sprain
Reproductive issues (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) — Clogged milk duct, irregular menses, mood swings with menstruation,
Eye infection (Eye disorders) | 1 (1) | 4 (7) | 0 (0) — Eye infection or pink eye
Dermatologic issues (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (4) — Mole removed with stitches, skin breakout, cyst on head
Ear infection (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Optic neuritis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain due to wisdom teeth extraction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Muffled hearing (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes